CLINICAL TRIAL: NCT06618794
Title: Recovery Legal Care Clinical Trial
Acronym: HVIP-MLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); U.S. Department of Justice (U.S. Federal Agency); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB24-0491; 4UH3HD111325-02 (NIH); P50MD017349 (NIH)
Record Dates: First submitted 2024-03-06; First posted 2024-10-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Firearm Injury; Economic Problems; Injury Traumatic; Racism, Systemic
Keywords: Firearm injury; Community violence; Medical-Legal Partnership; Systemic racism; Structural violence; Civil law attorneys; Health-Harming Legal Needs; Hospital-Based Violence Intervention Program
MeSH Terms: conditions — Wounds and Injuries; Systemic Racism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVIP-MLP (Experimental): This arm includes patients receiving usual care and also support from Recovery Legal Care (HVIP+MLP)
  Interventions: Other: Recovery Legal Care; Other: HVIP Standard of Care
- HVIP (Active Comparator): This arm includes patients receiving usual care (HVIP only).
  Interventions: Other: HVIP Standard of Care

INTERVENTIONS:
Other: Recovery Legal Care — These patients will receive support from our HVIP standard of care (Violence Recovery Program) plus our Medical Legal Partnership (Recovery Legal Care) for additional legal support to address health-harming legal needs and public benefits.
  Other Names: Civil Law Attorney Support; Public Benefits Attorney Support; Legal Aid Chicago Support
  Arms: HVIP-MLP
Other: HVIP Standard of Care — These patients will receive HVIP standard of care (Violence Recovery Program Support)
  Other Names: HVIP - Violence Recovery Program

SUMMARY:
Hospital-Based Violence Intervention Programs (HVIPs) affiliated with trauma centers in the US often focus on individual behavior modification for reduction in re-victimization. There is a lack of reproducible evidence that has demonstrated effectiveness, given the exclusion of addressing inequities in the Social and Structural Determinants of Health (SSDOH), often the root causes of violent injury and preventable homicide. The study investigators created a Medical Legal Partnership (MLP) to partner with an existing HVIP. This novel program offers beside legal assistance to address the SSDOH. The purpose of this study is to evaluate the effectiveness of the HVIP-MLP program in improving violence-related outcomes, legal needs, health-related quality of life, PTSD symptoms, and perceived stress.

DETAILED DESCRIPTION:
National trauma center verification relies on a commitment to injury prevention efforts, including prevention of community-level violence. Hospital-Based Violence Recovery Programs (HVIPs) have expanded across the country as extensions of level I and II trauma centers to address trauma recidivism with individual behavioral modification during the "teachable moment." There is little evidence that has demonstrated consistent effectiveness of this approach. One possible reason is the difficulty for community-based violence prevention specialists from HVIP programs to address the larger inequities in the Structural and Social Determinants of Health (SSDOH) that lead to violence through. Medical-Legal Partnership is one approach that has demonstrated evidence and success in improving health outcomes and reducing health-harming legal needs of patients, by connecting legal experts to medical experts for holistic care. This has yet to be done for trauma patients and has, to our knowledge, not been incorporated into any HVIP approach thus far. This clinical trial will evaluate the effectiveness of the HVIP-MLP model to address legal needs rooted in the SSDOH and improve violence-related outcomes. As secondary objectives, it will also evaluate whether the HVIP-MLP model can improve health-related quality of life, PTSD symptoms, and perceived stress among study participants. This novel HVIP-MLP approach has the potential to broadly impact the HVIP model to include an MLP component to all trauma centers for verification to support patients, families and providers alike in this important public health work.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for a violent injury at the University of Chicago Trauma Center
* Ages 14-64 years
* Able to provide informed consent (18 years and older) or assent (14-17 years)

Inclusion of women and minorities: This research proposal includes women and ethnic minorities. Patient participants will be primarily non-Hispanic Black or Hispanic race and ethnicity. The study expects participants to be proportional to the population-wide estimates for the South Side community. The majority will be low-income with variable functional health literacy. These characteristics are representative of the target population and describe the population most likely to benefit from the proposed study. Youth stakeholder participants will be multi-ethnic and racially diverse.

Inclusion of children: This study will include children ages 14-17 years old, based on Illinois state labor laws for child employment, as well as the ages of youth who are primarily treated for penetrating injury at the UCMC trauma center. This age is also a pragmatic cutoff for children providing meaningful input on community and healthcare solutions to violence.

Exclusion Criteria:

* Diagnosis of severe mental illness (i.e., psychotic disorder, schizophrenia, suicidality)
* Unable to provide informed consent due to mental status
* Prior receipt of legal services at UCMC within the past year
* Currently imprisoned or incarcerated
* Residing at an Indiana address.

Ages: 14 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Firearm victimization and aggression | Baseline, 3 months, 6 months, 12 months, 18 months
  The adapted Conflict Tactics Scale 2 (CTS2) measures behaviors related to firearm victimization and aggression over the past 3 months.

SECONDARY OUTCOMES:
Legal needs self-efficacy | Baseline, 3 months, 6 months, 12 months, 18 months
  The adapted Bandura Self-Efficacy Scale measures belief in one's ability to have legal needs addressed.
Health-related quality of life | Baseline, 3 months, 6 months, 12 months, 18 months
  The SF-12 Health Survey measures both physical and mental health domains of health-related quality of life.
Post-Traumatic Stress Disorder (PTSD) Symptoms | Baseline, 3 months, 6 months, 12 months, 18 months
  The PCL-5 measures symptoms of PTSD.
Stress | Baseline, 3 months, 6 months, 12 months, 18 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) scale measures self-reported psychological stress.

CONTACTS AND LOCATIONS:
Overall Officials: TANYA L ZAKRISON, MD, MPH, Principal Investigator — University of Chicago; ELIZABETH L TUNG, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this project will be shared with the Community Firearm Violence Prevention (CFVP) Network at the University of Michigan as part of a data sharing agreement stipulated under the UG3/UH3 award funding this research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available at the conclusion of data collection (11/1/2026) and will last for 5 years (10/31/2031).
Access Criteria: Data will be shared with trained and credentialed analysts from the CFVP team. They will be able to access de-identified survey data through an encrypted portal.

REFERENCES:
- See also: Program/intervention website — https://www.recoverylegal.uchicago.edu